CLINICAL TRIAL: NCT05637411
Title: GeoHealth: Geographic Information System for Health Management and Clinical, Epidemiological and Translational Research
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario Virgen Macarena (Other)
Responsible Party: Principal Investigator, Alberto Moreno Conde, PHD Alberto Moreno Conde, Hospital Universitario Virgen Macarena
Other Study IDs: PI19/01092
Record Dates: First submitted 2022-08-01; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Asthma; Allergy; Heart Diseases; Obesity; Rheumatic Diseases
MeSH Terms: conditions — Asthma; Hypersensitivity; Heart Diseases; Obesity; Rheumatic Diseases | interventions — Predictive Learning Models

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: The clinical data, socioeconomical data and environmental exposure data from 800.000 asthmatic patients attended in our region from 2007 to 2021 will be analysed to train and validate a risk predictive model for exacerbation (defined as emergency visits)
  Interventions: Other: Predictive model
- Prospective cohort: The same inclusion/exclusion criteria were applied prospectively. This is an external validation cohort.
  Interventions: Other: Predictive model

INTERVENTIONS:
Other: Predictive model — We will define and validate predictive models of risk of exacerbations in asthmatic patients

SUMMARY:
The objective of the project is to develop a potentially marketable system for clinical, epidemiological and translational research capable of associating contextual variables and geospatial data with clinical patient information. The GeoHealth system will include a section to perform exploratory analysis that will help identify risk factors to optimize clinical decision making. The system will be used in a study of the influence of environmental factors in more than 800,000 asthmatic patients in the region of Andalucía, Spain. The results of this study will help to develop predictive models of risk of exacerbation in asthma patients. Currently, disease management guidelines state that asthma control has two components: current disease control and future risk of exacerbations. These two components are key when assessing disease management, following a stepwise model that seeks to improve current control and minimize future risk. However, although the current control of the disease is defined and has established methodologies for its measurement (Asthma Control Test -ACT- and Asthma Control Questionnaire -ACQ-), the risk of suffering exacerbations is not yet a measurable component.

Therefore, these predictive models could help in professional decision making for asthmatic patients.

The predictive models will be validated prospectively and implemented in a decision support system for the management of asthmatic patients.

DETAILED DESCRIPTION:
The GeoHealth system will be designed as a modular platform that will allow communication to import patient data from EHR systems and research platforms through the ISO13606 and CDISC ODM standards. Furthermore, integrations will be made with the Andalusian HCE (Diraya) systems and the REDCap and OpenClinica clinical trial management systems.

GeoHealth integrates a set of heterogeneous open data sources, allowing a visualization, on the same map, of the clinical and contextual data of each patient based on their usual location (Census region of their home) and the desired date of the study. The data integrated into the system provide demographic information and the environmental conditions associated with the location of the patient.

The system has a module that perform analysis that can range from simple correlations between variables to other more complex analyzes such as clustering analysis, linear and logistic regressions and others.

Once the models that will be applied in decision-making have been determined, a study will be carried out on the degree of alignment between the recommendations established by the models and the clinical decision adopted by the professionals. The study will be performed during a period of 12 months in patients treated in the clinical centers that participate in this project.

The data come from different sources and all have been integrated into the same representation system. Using the free mapping system "OpenStreetMap" and the "Plotly" Python library, both the demographic data of the patients and their contextual variables are represented in a Dashboard, containing a single map.

The system offers the possibility to deploy different heat-maps using different regions (Census Regions, Postal Code Regions and Health Districts) and different demographic variables for each type of region (Population density, percentage of males and females, average incomes…etc.). Moreover, it is possible to choose between the different regions of Andalucía and a range of dates for the environmental (Pollution, pollen and meteorological data) and patient's data. Other places locations are deployed on the map as hospitals, clinics, roads and parks.

The system provides an advance in the deployment, observation and analysis for the health sector. It allows clinical researchers to understand better how the patient is affected by his environment and perform analysis to discover patterns in the data.

Other systems such as Transmart or i2b2, enable sharing, integration, standardization, and analysis of heterogeneous data from healthcare and translational research. GeoHealth has been presented as a possible extension of these two platforms helping them to incorporate the possibility to include geospatial data in the analysis.

Moreover, the system is going to be used and tested in two projects than aim to analyze the prevalence of asthmatic patients in the Macarena Hospital's area (Sevilla, Spain) and another in the region of Andalucía (Spain) where more than 800.000 patients will be analyzed.

It has been demonstrated how decisive the patient's environment is in the development of many diseases. GeoHealth has been presented as a platform that allows clinical researchers in the observation and analysis task to understand better how the environment affect them.

Moreover, the performed extraction, processing and integration of the open-data in the system and the intuitive deployment on a single map allow researchers to save time and access advanced analysis techniques that can be performed without the knowledge necessary to develop the algorithms that form them.

All these aspects make GeoHealth an innovative platform with a potential impact on the development of clinical studies related to the location and environment of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with bornchial asthma.

Exclusion Criteria:

* Women who are pregnant, breastfeeding or want to become pregnant during the duration of the study.
* Subjects with malignant disease, uncontrolled risk factors or any pathology that compromises the safety of the study.
* Subjects with problems that limit their ability to cooperate.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Our population is composed of patients with bornchial asthma.
Sampling Method: Probability Sample
Enrollment: 214 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Exacerbations | 1 year
  Measured by the number of times the patient goes to the emergency room or uses rescue medication and/or cycles of oral corticosteroids.

SECONDARY OUTCOMES:
Asthma control | 1 year
  Asthma control, obtained through the Asthma Control Test.
Quality-adjusted life year | 1 year
  To calculate this index, the EuroQol-5D quality of life questionnaire will be administered at baseline, three and six months into the study. The EQ-5D describes health status with five dimensions (mobility, self-care, activities of daily living, pain/discomfort, and anxiety/depression), each of which is defined with three levels of severity. It also consists of a millimetered Visual Analog Scale (VAS) on which the subject must score his or her health status on the day of the survey, with the extremes of the scale being the worst imaginable health status (0) and the best imaginable health status (100).
Respiratory function | 1 year
  Several pulmonary function tests will be carried out. These tests will include spirometry (FEV1, FVC, FEV1/FVC ratio, PC20, PD15, Fractional exhaled nitric oxide)
Immune response | 1 year
  IgE test, lymphocite count
Treatment adherence | 1 year
  estimated through dispensations

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Moreno, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Alberto Moreno Conde, Seville, Spain

IPD SHARING:
Plan to Share IPD: No